CLINICAL TRIAL: NCT04302818
Title: SKOLKONTAKT - Social Skills Training in a School Setting, a Randomized Controlled Pilot
Brief Title: SKOLKONTAKT - Social Skills Training in a School Setting
Acronym: SKOLKONTAKT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Marcus och Amalia Wallenbergs minnesfond (Unknown)
Responsible Party: Principal Investigator, Sven Bölte, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKOLKONTAKT
Record Dates: First submitted 2020-02-12; First posted 2020-03-10 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Anxiety; Depression
Keywords: Social skills group training; School-based intervention; Evidenced-based intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Teacher-assessors are blinded pre-, post, and follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social skills group training SKOLKONTAKT (Experimental): Manualised social skills group training.
  Interventions: Behavioral: SKOLKONTAKT
- Active control comparison group (Active Comparator): Social activities in a group setting.
  Interventions: Behavioral: Social activity group

INTERVENTIONS:
Behavioral: SKOLKONTAKT — N=21 participants are offered manualized and structured group training SKOLKONTAKT. The intervention includes 12 weeks, 3 sessions (50 minutes) per week.
  Other Names: SKOLKONTAKT Social skills training; SKOLKONTAKT Social skills group training; SKOLKONTAKT School-based social skills training
  Arms: Social skills group training SKOLKONTAKT
Behavioral: Social activity group — N=21 participants. The active comparison group includes 12 weeks, 3 sessions (50 minutes) per week. Sessions will include socially oriented activities such as board games, sports or baking as well as a recommended, general agenda.
  Arms: Active control comparison group

SUMMARY:
The study investigates the behavioral effects of an adapted manual-based social skills training program (SKOLKONTAKT) for the mainstream education plan delivered by school personnel, with pupils (15-20 years) with social-communication needs; either formally diagnosed (i.e. autism spectrum disorders or ADHD) or teacher-reported subclinical difficulties. N=40 are recruited from a community school in the Stockholm area (Sweden).

DETAILED DESCRIPTION:
So far, research has failed to consider the effectiveness of social skills training in school settings, and has instead focused on clinical or laboratory settings. This approach presents an interesting paradox given that the primary goal of social skills training is to affect change in the child's behavior in everyday life including school. Research undertaken in authentic everyday environments is not only more likely to result in real world outcomes for children and adolescents with ASD and ADHD, but greater utility in guiding models of service delivery. The objective of the current line of research is to adapt and evaluate methods originally designed to support children and adolescents with ASD and ADHD in clinical settings ("KONTAKT"), to be feasible and effective in school settings, that can be conducted by school personnel, and are are applicable to children with autistic and inattentive, hyperactive-impulsive disorders, as well as other less defined special social needs ("SKOLKONTAKT").

ELIGIBILITY:
Inclusion Criteria:

* Formally diagnosed autism spectrum disorder
* Formally diagnosed attention deficit hyperactivity disorder
* Teacher-reported subclinical social-communication special needs

Exclusion Criteria:

* Severe psychiatric comorbidity that challenges administration of the group-intervention, including but not limited to severe oppositional defiant disorder
* Severe psychiatric comorbidity that makes the participant to vulnerable to participate in the group-intervention, including but not limited to suicidality, severe depression

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Social Skills Group Questionnaire (SSGQ) | Change in score from baseline after 12 weeks of social skills training and at 3 months follow-up. Total time frame 6 months.
  Social skills (parent-, self- and (blinded) teacher-reported), higher score indicating improvement in skills

SECONDARY OUTCOMES:
Social Responsiveness Scale-2 (SRS-ll) | Change in score from baseline immediately after the intervention (12-13 weeks after baseline) and at 3 months follow-up (24-25 weeks after baseline). Total time frame 6 months.
  Autistic symptoms (parent-reported), decrease in scores indicating less clinical symptoms.
KIDSCREEN-27 (short version) | Change in score from baseline immediately after the intervention (12-13 weeks after baseline) and at 3 months follow-up (24-25 weeks after baseline).Total time frame 6 months.
  Health-related Quality of Life (self-reported).
Worlds Health Organisation Disability Assessment Schedule 2.0 (WHODAS 2.0) | Change in score from baseline immediately after the intervention (12-13 weeks after baseline) and at 3 months follow-up (24-25 weeks after baseline). Total time frame 6 months.
  Daily functioning as affected by functional disability (parent-reported).
Conners 3-F | Change in score from baseline immediately after the intervention (12-13 weeks after baseline) and at 3 months follow-up (24-25 weeks after baseline). Total time frame 6 months.
  ADHD-related symptoms (parent-reported), decrease in scores indicating less clinical symptoms.
Negative Effects Questionnaire (NEQ) | Change from baseline immediately after the intervention. Total time frame 3 months.
  Record of adverse events during intervention (parent-reported).
Goal Attainment Scaling (GAS) | Change in score from baseline immediately after the intervention (12-13 weeks after baseline). Total time frame 3 months.
  Personalised goal-setting (self-reported). Goal attaingment reported on a five-point scale, where higher score indicates better outcome.

OTHER OUTCOMES:
Pre-assessment questionnaire | At baseline.
  Expectations and person characteristics (parent and participant reported together) reported in a qualitative queastionnaire.
Evaluation questionnaire | Reported immediately after the intervention.
  Qualitative questionnaire for intervention evaluation (parent and participant reported together)
Evaluation questionnaire (school-staff) | Reported immediately after the intervention.
  Qualitative questionnaire for intervention evaluation (school-staff reported)
Evaluation questionnaire (principal) | Reported immediately after the intervention.
  Qualitative questionnaire for intervention evaluation (school principal-reported)
School grade | Change in score from baseline immediately after the intervention. Total time frame 3 months.
  Percent of grades indicating typical progress in subjects (teacher-reported)
School attendance | Change in score from baseline immediately after the intervention. Total time frame 3 months.
  Percent of school attendance (teacher-reported)
Attendance in intervention-group | Summary score of attended sessions. Scored immediately following every session of the intervention (3 sessions/week; 12 weeks). Total time frame 3 months.
  Number of sessions attended by participant (group-leader reported)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Bölte, Professor, Principal Investigator — CAP Research center, Karolinska Institutet
Locations (1):
- CAP Research Center, Center of Neurodevelopmental disorders at Karolinska Institutet (KIND), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choque Olsson N, Rautio D, Asztalos J, Stoetzer U, Bolte S. Social skills group training in high-functioning autism: A qualitative responder study. Autism. 2016 Nov;20(8):995-1010. doi: 10.1177/1362361315621885. Epub 2016 Feb 24. PMID 26912485
- [Background] Choque Olsson N, Flygare O, Coco C, Gorling A, Rade A, Chen Q, Lindstedt K, Berggren S, Serlachius E, Jonsson U, Tammimies K, Kjellin L, Bolte S. Social Skills Training for Children and Adolescents With Autism Spectrum Disorder: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2017 Jul;56(7):585-592. doi: 10.1016/j.jaac.2017.05.001. Epub 2017 May 10. PMID 28647010
- [Background] Jonsson U, Olsson NC, Coco C, Gorling A, Flygare O, Rade A, Chen Q, Berggren S, Tammimies K, Bolte S. Long-term social skills group training for children and adolescents with autism spectrum disorder: a randomized controlled trial. Eur Child Adolesc Psychiatry. 2019 Feb;28(2):189-201. doi: 10.1007/s00787-018-1161-9. Epub 2018 May 10. PMID 29748736
- See also: Homepage KIND. — http://ki.se/kind/center-of-neurodevelopmental-disorders-at-karolinska-institutet-kind